CLINICAL TRIAL: NCT05701839
Title: The Effect of Two Different Airway Management on Oxygenation During Deep Sedation in Patients Undergoing Hysteroscopy, Based on Oxygen Reserve Index Monitoring
Brief Title: Airway Management During Deep Sedation in Hysteroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XJTU1AF2022LSK-402
Record Dates: First submitted 2022-12-28; First posted 2023-01-27 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-10

CONDITIONS: Deep Sedation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- face mask airway management without oxygen reserve index monitoring (Experimental): Participants inhale oxygen through face mask at a flow rate of 5 L/min and will be monitored with oxygen saturation.
  Interventions: Procedure: face mask ventilation; Device: oxygen saturation monitoring
- face mask airway management with oxygen reserve index monitoring (Experimental): Participants inhale oxygen through face mask at a flow rate of 5 L/min and will be monitored with oxygen reserve index.
  Interventions: Procedure: face mask ventilation; Device: oxygen reserve index monitoring
- nasopharyngeal tube airway management without oxygen reserve index monitoring (Experimental): Participants inhale oxygen through face mask before induction and through nasopharyngeal tube after consciousness disappear at a flow rate of 5 L/min and will be monitored with oxygen saturation.
  Interventions: Procedure: nasopharyngeal tube ventilation; Device: oxygen saturation monitoring
- nasopharyngeal tube airway management with oxygen reserve index monitoring (Experimental): Participants inhale oxygen through face mask before induction and through nasopharyngeal tube after consciousness disappear at a flow rate of 5 L/min and will be monitored with oxygen reserve index.
  Interventions: Procedure: nasopharyngeal tube ventilation; Device: oxygen reserve index monitoring

INTERVENTIONS:
Procedure: face mask ventilation — In participants with face mask ventilation, oxygen inhaled through face mask at a flow rate of 5 L/min.
  Arms: face mask airway management with oxygen reserve index monitoring; face mask airway management without oxygen reserve index monitoring
Procedure: nasopharyngeal tube ventilation — In participants with nasopharyngeal tube ventilation, oxygen inhaled through face mask before induction and through nasopharyngeal tube after consciousness disappear at a flow rate of 5 L/min.
  Arms: nasopharyngeal tube airway management with oxygen reserve index monitoring; nasopharyngeal tube airway management without oxygen reserve index monitoring
Device: oxygen saturation monitoring — In participants with oxygen saturation monitoring, assist ventilation through face mask will be performed when oxygen saturation drops to 95%, it lasts for another 10 seconds when oxygen saturation restores to 100%.
  Arms: face mask airway management without oxygen reserve index monitoring; nasopharyngeal tube airway management without oxygen reserve index monitoring
Device: oxygen reserve index monitoring — In participants with oxygen reserve index monitoring, assist ventilation through face mask will be performed when oxygen reserve index drops to 0.1, it lasts for another 10 seconds when oxygen reserve index restores to 0.1.
  Arms: face mask airway management with oxygen reserve index monitoring; nasopharyngeal tube airway management with oxygen reserve index monitoring

SUMMARY:
Hysteroscopy is used to examine and treat uterine diseases. Because of severe pain due to uterine distention and cervical dilatation, deep sedation usually be provided during this procedure. Respiratory depression and upper airway obstruction are main respiratory complications during deep sedation. Face mask and nasopharyngeal airway are main airway management during deep sedation. Oxygen reserve index is a non-invasive parameter, it reflects the moderate hyperoxia statues. In this study, investigators compare the effect of face mask and nasopharyngeal airway management on oxygenation during deep sedation in participants undergoing hysteroscopy. Investigators also investigate whether oxygen reserve index monitoring reduce the incidence of hypoxemia.

DETAILED DESCRIPTION:
Randomization:

Participants are divided into four groups: face mask airway management without oxygen reserve index (ORi) monitoring group (FM-ORi group), face mask airway management with ORi monitoring group (FM+ORi group), nasopharyngeal tube airway management without ORi monitoring group (NT-ORi group), nasopharyngeal tube with ORi monitoring group (NT+ORi group).

Deep sedation process:

Participants fasting solid and liquid for 8 and 4 hours respectively. Electrocardiogram (ECG), oxygen saturation (SpO2), blood pressure (BP) and bispectral index (BIS) were monitored. Sufentanil 5 μg injected for 30 seconds, followed by target-control infusion of propofol (plasma target concentration 3-6 ug/ml) to maintain BIS between 50-70. Criteria for deep sedation: participants have purposeful response after repeated and/or painful stimulation, there is minimal effect on hemodynamic stability.

Airway management:

In FM-ORi and FM+ORi group, participants spontaneous inhaled oxygen through face mask at a flow rate of 5 L/min. in FM-ORi group, assist ventilation through face mask was performed when SpO2 dropped to 95%, it lasted for another 10 seconds when SpO2 restored to 100%. In FM+ORi group, assist ventilation through face mask was performed when ORi dropped to 0.1, it lasted for another 10 seconds when ORi restored to 0.1.

In NT-ORi and NT+ORi group, participants spontaneous inhaled oxygen through face mask before induction and through nasopharyngeal tube after consciousness disappear at a flow rate of 5 L/min. in NT-ORi group, assist ventilation through face mask was performed when SpO2 dropped to 95%, it lasted for another 10 seconds when SpO2 restored to 100%. In NT+ORi group, assist ventilation through face mask was performed when ORi dropped to 0.1, it lasted for another 10 seconds when ORI restored to 0.1.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18-60 years old
* Scheduled for hysteroscopy
* Predict operation duration more than 10 minutes

Exclusion Criteria:

* Participants refuse
* Predict the presence of difficult airway
* Combined with obstructive sleep apnea syndrome
* Combined with upper respiratory tract infection, and/or pulmonary inflammation
* Combined with chronic obstructive pulmonary disease
* Combined with asthma
* Body mass index (BMI) >30 kg/m2
* Coagulation dysfunction, and/or undergo anticoagulant therapy
* Nasal deformity
* Pregnancy, positive urine pregnancy test

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of low oxygen saturation | Procedure (from anesthesia induction to anesthesia recovery)
  oxygen saturation less than 95% last for at least 10 seconds

SECONDARY OUTCOMES:
Total duration of assist ventilation | Procedure (from anesthesia induction to anesthesia recovery)
  cumulative assist ventilation time during sedation in one patient
The lowest oxygen saturation | Procedure (from anesthesia induction to anesthesia recovery)
  the lowest oxygen saturation during sedation

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Guan, MD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Investigators have no plan to make individual participant data available to other researchers